CLINICAL TRIAL: NCT00287079
Title: A Prospective, Open Label, Multi-centre Study Exploring the Use of Subcutaneous (sc) 44 Microgram Interferon (IFN) Beta - 1a (Rebif®) Once a Week (qw) in Subjects With Clinically Isolated Syndrome (CIS)
Brief Title: A Prospective Study Looking at the Use of Rebif® in Subjects With Clinically Isolated Syndrome
Acronym: CIS-ON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Serono Canada Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 26222
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Clinically Isolated Syndrome
MeSH Terms: interventions — Interferon beta-1a

ARMS (2):
- Rebif® (Experimental)
  Interventions: Drug: Rebif®
- No Treatment (Other)
  Interventions: Other: No Treatment

INTERVENTIONS:
Drug: Rebif® — 44 microgram (mcg) IFN beta-1a sc once a week (qw) for 96 weeks
  Arms: Rebif®
Other: No Treatment — No treatment for 96 weeks
  Arms: No Treatment

SUMMARY:
The primary objective of this initiative is to assess the effectiveness of subcutaneous (sc) interferon (IFN) beta - 1a, (Rebif®), versus No Treatment in delaying the conversion to Clinically Definite Multiple Sclerosis (CDMS) - as defined by the occurrence of a second exacerbation - over 96 weeks in subjects that present with Clinically Isolated Syndrome (CIS) accompanied by an abnormal magnetic resonance imaging (MRI). The secondary objectives are to:

* Assess the effectiveness of sc IFN beta - 1a (Rebif®) therapy in reducing the proportion of patients with CIS converting to CDMS
* Assess the safety of sc IFN beta - 1a (Rebif®) in the patients with CIS

ELIGIBILITY:
Inclusion Criteria:

* Subject must have experienced a first clinical episode suggestive of demyelinating disease
* Subject must present with an abnormal MRI displaying at least 3 T2 weighted hyperintense lesions typical of multiple sclerosis (MS)
* Subject must be greater than or equal to 18 years old
* Subject must have had onset of the clinical attack within the last 120 days
* Subject must give written informed consent
* Female subjects must be neither pregnant nor breast feeding, and must not be of child-bearing potential as defined by either:
* Being post-menopausal or surgically sterile
* Using hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study

Subjects electing treatment:

* Subject must be eligible for Interferon-beta 1-a therapy

Exclusion Criteria:

* Subject has evidence of other neurological diseases that could explain his/her symptomatology
* Subject is pregnant or in lactation
* Subject suffers from an intercurrent autoimmune disease
* Subject suffers from major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the procedures required by this study
* Subject has received immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporine, methotrexate, azathioprine, linomide, mitoxantrone, teriflunomide, natalizumab, laquinimod, campath), within 12 months of study day 1

Subjects electing treatment:

* Subject has inadequate liver function, defined by total bilirubin, aspartate transaminase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal values
* Subject has inadequate bone marrow reserve, defined as white blood cell count less than 0.5 times the lower limit of normal
* Subject has a known allergy to IFN or any of the excipients of the drug product

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — EMD Serono Canada Inc.
Locations (1):
- Canadian Medical Information Office, Windsor, Barrie, Hamilton, Mississauga, Ontario, Canada

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebif 44 Mcg: Rebif was administered subcutaneously (sc) at a dose of 44 microgram (mcg) once weekly.
- No Treatment: Participants in this group did not receive any treatment.
Period: Overall Study
Arm/Group | Rebif 44 Mcg | No Treatment
Started | 32 | 3
Completed | 10 | 2
Not Completed | 22 | 1
Not completed — Qualifying relapse | 12 | 1
Not completed — Non-qualifying relapse | 1 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif 44 Mcg | No Treatment | Total
Number analyzed (Participants) | 32 | 3 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.30 (9.68) | 35.30 (13.32) | 35.80 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 3 | 22
  Male | 13 | 0 | 13

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Converted to Clinical Definite Multiple Sclerosis (CDMS)
Description: CDMS was defined as the occurrence of a second exacerbation over 96 weeks in participants who presented with CIS accompanied by an abnormal MRI scan.
Time Frame: Up to Week 96
Population: Intent-to-treat (ITT) population: All participants in Treatment group who received at least 1 dose of Rebif® and all participants in observational group who had at least 1 post-baseline visit were included in ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Rebif 44 Mcg | No Treatment
Number analyzed (Participants) | 32 | 3
Percentage of participants | 37.5 | 33.3

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition.
Time Frame: Up to Week 96
Population: Intent-to-treat (ITT) population: All participants in Treatment group who received at least 1 dose of Rebif® and all participants in observational group who had at least 1 post-baseline visit were included in ITT population. Adverse events were not captured for "No Treatment" group.
Measure: Number; unit: percentage of participants
Arm/Group | Rebif 44 Mcg | No Treatment
Number analyzed (Participants) | 32 | 0
percentage of participants | 100 |

3. Primary Outcome: Time in Month to Clinical Definite Multiple Sclerosis (CDMS) From Kaplan-Meier Estimates
Description: CDMS was defined by the occurrence of a second exacerbation or relapse over 96 weeks in participants who presented with Clinically Isolated Syndrome (CIS) accompanied by an abnormal Magnetic Resonance Imaging (MRI) scan. Time was calculated from the date of the stabilization of the baseline CIS episode to the qualifying relapse for the CDMS.
Time Frame: Up to Week 96
Population: Intent-to-treat (ITT) population: All participants in Treatment group who received at least 1 dose of Rebif® and all participants in observational group who had at least 1 post-baseline visit were included in ITT population. Two participants had negative time from stabilization and CDMS relapse and were excluded from the Kaplan-Meier analysis.
Measure: Mean (Standard Error); unit: Month
Arm/Group | Rebif 44 Mcg | No Treatment
Number analyzed (Participants) | 30 | 3
Month | 15.6 (1.23) | 17.0 (NA) — Standard Error not analyzed due to limited number of participants

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: AE: any untoward medical occurrence in form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered. AE were not captured for "No Treatment" group.
Arm/Group | Rebif 44 Mcg | No Treatment
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/0
Other Adverse Events (participants affected / at risk) | 32/32 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif 44 Mcg (N=32) | No Treatment (N=0)
Mild Leucopenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif 44 Mcg (N=32) | No Treatment (N=0)
Visual Disturbance (Eye disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 10 | 0
Stomach Discomfort (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Chills (General disorders) | 16 | 0
Fatigue (General disorders) | 17 | 0
Influenza like illness (General disorders) | 7 | 0
Injection site bruising (General disorders) | 3 | 0
Injection site discomfort (General disorders) | 2 | 0
Injection site erythema (General disorders) | 5 | 0
Injection site irritation (General disorders) | 4 | 0
Injection site pain (General disorders) | 3 | 0
Pain (General disorders) | 12 | 0
Pyrexia (General disorders) | 4 | 0
Influenza (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 9 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Balance Disorder (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysaesthesia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 23 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 0
Paraesthesia (Nervous system disorders) | 5 | 0
Depression (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other